CLINICAL TRIAL: NCT01898845
Title: A Phase I Study of LEE011 in Asian Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of LEE011 in Asian Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X1101
Record Dates: First submitted 2013-07-01; First posted 2013-07-12 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-07

CONDITIONS: Advanced Solid Tumors
Keywords: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LEE011 (Experimental): LEE011
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011

SUMMARY:
This study will evaluate safety and tolerability to estimate the MTD and/or recommended dose for expansion.

DETAILED DESCRIPTION:
This is a multi-center, open label, dose finding, phase I study of oral single agent LEE011, administered once daily.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a histologically confirmed diagnosis of a solid tumor
* ECOG PS <2
* Good organ function at screening visit
* A sufficient interval mast have elapsed between the last dose of prior anti-cancer therapy

Exclusion Criteria:

* Impairment of GI function
* Patients with concurrent severe and/or uncontrolled concurrent medical conditions
* Known diagnosis of HIV or active viral hepatitis
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | First cycle (28 days)
Maximum tolerated dose (MTD) and/or recomended dose (RD) | First cycle (28 days)

SECONDARY OUTCOMES:
Safety and Tolerability of LEE011 | from informed consent till 28 days after end of treatment
  Assessed by incidence, duration and severity of adverse events and serious adverse events; changes in clinical laboratory values, vital signs and ECGs; tolerability of study drug (dose interruption, dose reduction)
PK parameters of LEE011 | every week up to first 4 weeks, once a week in the subsequent 2 weeks
  Concentration of LEE011 and PK parameters (e.g. Cmax and AUC)
Best overall response | every 2 months until 28 days after end of treatment
  To assess preliminaly anti-tumor activity based on RECIST
Overall response rate | every 2 months until 28 days after end of treatment
  To assess preliminaly anti-tumor activity based on RECIST
Progression-free survival | every 2 months until 28 days after end of treatment
  To assess preliminaly anti-tumor activity based on RECIST
Disease control rate | every 2 months until 28 days after end of treatment
  To assess preliminaly anti-tumor activity based on RECIST
Duration of response | every 2 months until 28 days after end of treatment
  To assess preliminaly anti-tumor activity based on RECIST
Overall response | every 2 months until 28 days after end of treatment
  To assess preliminaly anti-tumor activity based on RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Chuo-ku, Tokyo

REFERENCES:
- [Result] Doi T, Hewes B, Kakizume T, Tajima T, Ishikawa N, Yamada Y. Phase I study of single-agent ribociclib in Japanese patients with advanced solid tumors. Cancer Sci. 2018 Jan;109(1):193-198. doi: 10.1111/cas.13428. Epub 2017 Nov 12. PMID 29059492
- [Derived] Ji Y, Yartsev V, Quinlan M, Serra P, Wang Y, Chakraborty A, Miller M. Justifying Ribociclib Dose in Patients with Advanced Breast Cancer with Renal Impairment Based on PK, Safety, and Efficacy Data: An Innovative Approach Integrating Data from a Dedicated Renal Impairment Study and Oncology Clinical Trials. Clin Pharmacokinet. 2023 Mar;62(3):493-504. doi: 10.1007/s40262-022-01206-2. Epub 2023 Feb 17. PMID 36800111
- See also: Results for CLEE011X1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14108